CLINICAL TRIAL: NCT05870397
Title: Optimal Recheck Time for Helicobacter Pylori Eradication: A Prospective, Single-center, Open-label, Randomized Controlled Trial
Brief Title: Optimal Recheck Time for Helicobacter Pylori Eradication: A Prospective Randomized Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-0184
Record Dates: First submitted 2023-05-04; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-04

CONDITIONS: Helicobacter Pylori Eradication

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a single-center, open-label, randomized controlled study in Zhejiang, China. Treatment-naive H. pylori-positive participants (n = 900) were randomly assigned to three groups in a 1:1:1 ratio with the same eradication regimen: amoxicillin 1000 mg, clarithromycin 500mg, rabeprazole 10mg, and colloidal bismuth 200 mg each given twice a day for 14 days. Urea breath tests were administered at different times after treatment: 4 to 6 weeks, 6 to 8 weeks, and 8 to 10 weeks, respectively, for different groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Recheck time is at 4 to 6 weeks after the eradication therapy (Placebo Comparator): All cases are administered the same eradication regimen: amoxicillin 1000 mg, clarithromycin 500mg, rabeprazole 10mg, and colloidal bismuth 200 mg each given twice a day for 14 days. Urea breath tests were administered at 4 to 6 weeks( as guildeline suggested) after the treatment.
  Interventions: Diagnostic Test: HY-IREXB plus carbon 13 breath detector do the breath urea test after eradication at different times
- Recheck time is at 6 to 8 weeks after eradication therapy (Active Comparator): All cases are administered the same eradication regimen: amoxicillin 1000 mg, clarithromycin 500mg, rabeprazole 10mg, and colloidal bismuth 200 mg each given twice a day for 14 days. Urea breath tests were administered at 6 to8 weeks after the treatment.
  Interventions: Diagnostic Test: HY-IREXB plus carbon 13 breath detector do the breath urea test after eradication at different times
- Recheck time is at 8 to 10 weeks after eradication therapy (Active Comparator): All cases are administered the same eradication regimen: amoxicillin 1000 mg, clarithromycin 500mg, rabeprazole 10mg, and colloidal bismuth 200 mg each given twice a day for 14 days. Urea breath tests were administered at 8 to 10 weeks after the treatment.
  Interventions: Diagnostic Test: HY-IREXB plus carbon 13 breath detector do the breath urea test after eradication at different times

INTERVENTIONS:
Diagnostic Test: HY-IREXB plus carbon 13 breath detector do the breath urea test after eradication at different times — Carbon 13 breath tests are generally performed 4-6 weeks after eradication therapy. The control group will perform breath urea test at 4-6 weeks after treatment. The experimental groups will perform the same test at different times after the same treatment, 6-8weeks and 8-10 weeks, respectively.

SUMMARY:
Although Urea breath test has been commonly used to recheck the efficiency of Helicobacter pylori eradication, there has been no randomized trials comparing the accuracy of Urea breath test results at different times after eradication. The investigators aim to assess the accuracy and influence factors of post-therapy test at different times and follow up the cut off samples to optimize the best time to recheck.

DETAILED DESCRIPTION:
The investigators plan to conduct a single-center, open-label, randomized controlled study in Zhejiang, China. Treatment-naive H. pylori-positive participants (n = 900) were randomly assigned to three groups in a 1:1:1 ratio with the same eradication regimen: amoxicillin 1000 mg, clarithromycin 500mg, rabeprazole 10mg, and colloidal bismuth 200 mg each given twice a day for 14 days. Urea breath tests were administered at different times after the treatment: 4 to 6 weeks, 6 to 8 weeks, and 8 to 10 weeks, respectively, for different groups.

ELIGIBILITY:
Inclusion Criteria:

* no history of helicobacter pylori treatment
* the diagnosis of H. pylori infection was confirmed by one or more of the following methodologies before treatment: gastric biopsy using histochemical staining, tissue culture, the 14C-urea breath test (UBT), and/or the 13C-UBT.

Exclusion Criteria:

* used antibiotics or bismuth within four weeks before inclusion or acid inhibitor use, including H2 receptor antagonist (H2RA), PPI or P-CAB use, within two weeks prior to inclusion.
* had an active peptic ulcer with complications such as hemorrhage, perforation, or obstruction.
* had a history of esophagectomy or gastrectomy.
* had an allergy to any study drug.
* had severe comorbidities or physical or mental diseases.
* were pregnant or breastfeeding.
* had a history of alcohol abuse or drug addiction.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2023-04-21 (Actual); Primary Completion 2024-04-21 (Estimated); Study Completion 2024-08-21 (Estimated)

PRIMARY OUTCOMES:
the eradication rate in each group (ITT analysis) | up to 4 months after eradication therapy
  According to the breath urea test, calculation the eradication rate in the three groups. ITT analysis, the number of negative breath test cases after treatment divided by the number of cases enrolled in eradication therapy.
the eradication rate in each group (PP analysis) | up to 4 months after eradication therapy
  According to the breath urea test, calculation the eradication rate in the three groups. PP analysis, the number of negative breath test cases after treatment divided by the number of cases finished the eradication therapy

SECONDARY OUTCOMES:
follow up of cut off cases | up to 4 months after eradication therapy.
  If the result of breath urea test is betwwen 2 to 6, it will be defined as cut off value. These cases will be collected and take further tests to make sure the real situation of helicobacter pylori infection.

CONTACTS AND LOCATIONS:
Overall Officials: Jianting Cai, MD, Study Chair — 2nd Affilicated Hosptal,School of Medicine,Zhejiang University,China
Locations (1):
- 2nd Affilicated Hosptal,School of Medicine,Zhejiang University,China, Hangzhou, Zhejiang, China